CLINICAL TRIAL: NCT07065500
Title: Mechanism and Effect of Novel Metabolites on Valvular Heart Disease（Hestia Study）
Brief Title: Mechanism and Effect of Novel Metabolites on Valvular Heart Disease
Acronym: Hestia
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Principle Investigator, Sun Yat-sen University
Other Study IDs: Hestia study
Record Dates: First submitted 2025-07-02; First posted 2025-07-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-03

CONDITIONS: Valvular Heart Disease
Keywords: novel metabolites; valvular heart disease; prognosis; Risk Factors
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical diagnosis of heart valve disease

SUMMARY:
Valvular heart disease (VHD) is a leading cause of loss of physical function, reduced quality of life and increased longevity.The epidemiology of VHD varies widely across the globe, with functional and degenerative diseases occurring predominantly in high-income countries and rheumatic heart disease occurring predominantly in low- and middle-income countries. The prevalence of valvular heart disease (VHD) is increasing globally due to improved survival and aging populations, poorly controlled by medications, with the majority of patients having to undergo surgical or interventional treatments.

It is therefore important to search for novel metabolites and conduct mechanistic studies on the effects of these metabolites on patients with heart valve disease.

In the Hestia study, the investigators looked for risk factors and mechanisms associated with the development and prognosis of VHD through long-term follow-up of VHD patients and metabolite testing of specimen tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender is not limited.
2. Clinical diagnosis of heart valve disease (including aortic stenosis, aortic valve closure insufficiency due to different etiologies, mitral stenosis, mitral valve closure insufficiency, pulmonic stenosis, pulmonic valve closure insufficiency, tricuspid stenosis and tricuspid closure insufficiency due to different etiologies )

Exclusion Criteria:

Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with valvular heart disease during hospitalization were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with All-cause mortality | 5 years

SECONDARY OUTCOMES:
Number of Participants with cardiovascular events | 5 years
Number of Participants with progression of valvular heart disease | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen Univerity, Guangzhou, Guangdong, China